CLINICAL TRIAL: NCT04354298
Title: Effects of Improvisational Dance on Cognition and Daily Function Among People With Parkinson Disease
Brief Title: Improvisational Dance for Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Lee Silverman Voice Training Global (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 201905089
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: dance; cognition; daily function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fall 2019 ID Class (Experimental): The ID group participated in a 12-week IMPROVment® intervention, which consists of weekly ID classes that progress according to a standardized method, from September 2019-December 2019.
  Interventions: Behavioral: Improvisational Dance Class
- Fall 2020 ID Class (Experimental): The ID group will participate in a 12-week IMPROVment® intervention, which consists of weekly ID classes that progress according to a standardized method, from September 2020-December 2020.
  Interventions: Behavioral: Improvisational Dance Class
- Control Group (No Intervention): Participants are pre- and post-tested 12-14 weeks apart after not having changed anything drastic in their daily life.

INTERVENTIONS:
Behavioral: Improvisational Dance Class — Hour long movement classes that meet weekly for 12 weeks.
  Arms: Fall 2019 ID Class; Fall 2020 ID Class

SUMMARY:
The long-term goal of this work is to maintain or improve daily function of people with PD by addressing cognition. The overall objective is to discover interventions that aid in cognitive functioning. The central hypothesis is that engagement in an improvisational dance (ID) class will benefit cognition among people with PD. Improvisational dance involves spontaneously generated movement, similar to how one moves in everyday life. The literature shows that ID classes positively impact motor impairments associated with PD, such as balance, gait, and functional mobility. Along with being physically demanding, ID requires the use and coordination of a number of cognitive capacities to properly execute movements. This type of activity challenges, and thus may strengthen, cognitive processes such as motor planning, decision making, flexible thinking, initiation, and execution, which may give people cognitive based strategies to be utilized in various aspects of daily life. By improving motor function and/or cognition, ID may also contribute to improved daily functioning, or the ability to perform and participate in daily activities. Despite these theoretical links, evidence for the effect of ID on cognition and overall daily function is limited. The current project objective is to address this gap and better understand the effects of ID for people with PD. Specifically, it will test the effect of IMPROVment®, a method of ID designed for people with PD, on cognition and daily function.

Participants' cognition will be assessed at baseline (T1) using the NIH Toolbox Cognitive Battery, the Alternate Uses Task, and the Weekly Calendar Planning Activity. Global cognition will be assessed using the Montreal Cognitive Assessment. They then will be randomly assigned to either the immediate intervention (ID) or waitlist-control (WC) group. The ID group will start the 12-week IMPROVment® intervention, which consists of weekly ID classes that progress according to a standardized method while the WC group will receive no intervention and continue with their regular daily routine and activity level. After 12 weeks, both groups will complete cognitive testing again (T2). Cognitive test scores will be compared across time points and between groups using a mixed model repeated measures ANOVA. The investigators hypothesize that IMPROVment® will have positive effects on the cognitive abilities of people with PD. Participants will also complete two questionnaires to assess daily function at T1 and T2: Older Americans Resources and Services Scale- Extended Version and PROMIS Satisfaction with Participation in Discretionary Social Activities. These scores will be compared similar to the above aim. The investigators hypothesize that IMPROVment® will have positive effects on daily function in people with PD.

Participant mood will be assessed in two different ways. The first being to investigate the immediate effect of participating in an IMPROVment® class on mood, fatigue, and anxiety. The investigators hypothesize that mood will positively improve from pre to post of each class. To assess this, participants will respond to a scale assessing mood, specifically sadness, nervousness, energy, and overall well-being before and after each class every week. The second measurement is to investigate the effect of IMPROVment® on anxiety, fatigue, and depression. The investigators hypothesize that IMPROVment® class will decrease feelings of depression for those with PD. All participants will fill out the Parkinson's Anxiety Scale, the Parkinson's Disease Fatigue Scale, and the Geriatric Depression Scale short form before and after participating in the 12-week IMPROVment® program.

Achievement of these aims will provide further support for the IMPROVment® method for people with PD experiencing cognitive deficits. The long-term impact will better cognition and daily functioning in people with PD, and thus enhanced everyday lives.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 years or older
* Parkinson Disease Diagnosis
* Hoehn-Yahr score between 1-3
* independently walk at least 3 meters
* cognitive ability to follow simple commands

Exclusion Criteria:

* Montreal Cognitive Assessment score less than or equal to 22
* diagnosis of other severe comorbidities
* contraindications to physical activity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Cognition (National Institute of Health Toolbox: Cognitive Battery) | Before and After the 12-week intervention
  A comprehensive, performance-based test comprised of motor, emotion, sensation, and cognition assessments. For the purpose of this study, the investigators will be using the cognitive battery to assess processes involved in learning and comprehension (i.e. thinking, remembering, problem-solving, judging). The battery consists of tasks involving the use of executive function, memory, attention, and language.
Change in Cognition (Alternate Uses Task) | Before and After the 12-week intervention
  A verbal test of divergent thinking where the participant is given the name of an object and must name as many uses of that object as possible in a 3-minute time period. This assessment measures verbal fluency, originality, flexibility, and elaboration.
Change in Functional Cognition (Weekly Calendar Planning Activity) | Before and After the 12-week intervention
  A performance-based measure that assesses an individual's level of executive function. The task involves entering a list of errands into a calendar while following rules, keeping track of time, and managing conflicts.
Change in Daily Performance (Older American Resources and Services Scale) | Before and After the 12-week intervention
  A self-report questionnaire-based assessment that assesses perceived performance in activities of daily living and instrumental activities of daily living by reporting the level of difficulty that they experience while completing the specific activity. Areas assessed include activities of daily living (walking, eating, dressing, grooming, getting in and out of bed, bathing, and toileting) and instrumental activities of daily living (using a telephone, traveling, shopping, preparing meals, housework, managing medication, and handling money). Higher scores are associated with increased daily performance.
Change in Daily Participation (PROMIS Satisfaction with Participation in Discretionary Social Activities) | Before and After the 12-week intervention
  A self-report questionnaire-based assessment that assesses satisfaction in ability to participate in activities of daily living and instrumental activities of daily in the past 7 days. Higher scores are associated with increased daily participation.
Change in Anxiety (Parkinson's Anxiety Scale) | Before and After the 12-week intervention
  A self-report measure of anxiety specifically for people with PD. It includes three subscales: persistent anxiety, episodic anxiety, and avoidance behavior, and scores for each section can be determined by summing the items in each subscale. The total score is a summation of the subscales, and higher scores indicate greater anxiety.
Change in Level of Fatigue (Parkinson's Disease Fatigue Scale) | Before and After the 12-week intervention
  A self-report measure assessing the presence of fatigue in people with PD. It focuses on the physical aspects of fatigue and their effect on activities and daily function. Item scores are averaged, with a score of >2.95 indicating presence of fatigue.
Change in Depressive Symptoms (Geriatric Depression Scale) | Before and After the 12-week intervention
  A self-report questionnaire assessing depression in older adults. Item scores are summed to yield a total score, and a score 5 ≥ warranting a follow up interview and a score greater than 10 almost always indicating depression.
Change in Overall Mood After Each Class (Visual Analog Scales) | Before and After each ID Class taken for 12-weeks.
  This consisted of four sliding scales (very sad to very happy; very calm to very nervous; very lively to very sluggish; overall well being: very poor to very well) on a 100mm line. A higher score on the very sad to very happy and overall well being scales indicated greater happiness and better overall well being while a lower score on the very calm to very nervous and lively to sluggish scale indicate more calmness and liveliness.

SECONDARY OUTCOMES:
Change in Motor Symptoms (Unified Parkinson Disease Rating Scale: Motor Battery) | Before and After the 12-week intervention
  A scale that is used to rate the severity of PD symptoms, and the motor scale focuses on the motor-related symptoms. Higher scores are associated with increased presence of motor symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- 4444 Forest Park Ave., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Participants consented to their data being shared with other researchers. Future students may use this data to draw further conclusions.

REFERENCES:
- [Background] Batson G, Hugenschmidt CE, Soriano CT. Verbal Auditory Cueing of Improvisational Dance: A Proposed Method for Training Agency in Parkinson's Disease. Front Neurol. 2016 Feb 17;7:15. doi: 10.3389/fneur.2016.00015. eCollection 2016. PMID 26925029
- [Background] Hashimoto H, Takabatake S, Miyaguchi H, Nakanishi H, Naitou Y. Effects of dance on motor functions, cognitive functions, and mental symptoms of Parkinson's disease: a quasi-randomized pilot trial. Complement Ther Med. 2015 Apr;23(2):210-9. doi: 10.1016/j.ctim.2015.01.010. Epub 2015 Jan 16. PMID 25847558
- [Background] McNeely ME, Duncan RP, Earhart GM. Impacts of dance on non-motor symptoms, participation, and quality of life in Parkinson disease and healthy older adults. Maturitas. 2015 Dec;82(4):336-41. doi: 10.1016/j.maturitas.2015.08.002. Epub 2015 Aug 12. PMID 26318265
- [Background] Soriano, C. T., & Batson, G. (2011). Dance-making for adults with Parkinson disease: one teacher's process of constructing a modern dance class. Research in Dance Education, 12(3), 323-337. doi: 10.1080/14647893.2011.614334

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT04354298/Prot_SAP_ICF_000.pdf